CLINICAL TRIAL: NCT02648594
Title: Efficacy Assessment of CT-guided Hook Wire Localization of Lung Nodes With Medical Device " Fil d'Ariane " Laurane médical Before Thoracoscopy- HARNO Trial
Brief Title: Efficacy Assessment of CT-guided Hook Wire Localization of Lung Nodes Before Thoracoscopy
Acronym: HARNO
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: A retrospective study has already been conducted on the same topic
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-A00958-41
Record Dates: First submitted 2015-12-23; First posted 2016-01-07 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Nodes, Lung
Keywords: lung; thoracoscopy; hook wire localization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention: Hook wire CT guided (Experimental): There is only one arm. When patient undergo surgery , the radiologist will place a CT-guided Hook wire in order to localize it in patient lung. The intervention consists to place a CT-guided hook wire in contact with the pulmonary nodule under local anesthesia.
  Then, the thoracoscopy will be realised. Then, the surgery piece will be examined to confirm if the node is in the surgery piece
  Interventions: Device: Hook wire CT guided

INTERVENTIONS:
Device: Hook wire CT guided — The intervention consist to place a CT-guided hook wire in lung patient

SUMMARY:
When patient presents a lung node, there is an important risk that this node was a tumor. For patients who have these nodes, the surgery is the best treatment. When the surgery is possible, the thoracoscopy may be more advantageous compared to thoracothomy (decrease of post surgery pains, decrease of recovery time and decrease of drugs consumption). Nevertheless, thoracoscopy needs specific materiels and nécessite un équipement spécifique and trained physicians.

Moreover, this technic needs that nodes was well localized. For this, radiologists use CT-guided hook wire localization of these lung nodes before surgery.

TThe hook wire laying is delicate. It can lead secondaries effects as pneumothorax, dislodgement of the hook wire before and after surgery. The success rate of hook wire fixation in lung near of the node is primary.

The main objective of our study is to assess the success rate localization of node in surgery piece, that is to verify if the hook wire have allowed to localize the lung node in surgery piece.

DETAILED DESCRIPTION:
For lung cancer patients, the best treatment remains the surgery when tumor is localized.

When patient presents a lung node, there is an important risk that this node was a tumor. For patients who have these nodes, the surgery is the best treatment. When the surgery is possible, the thoracoscopy may be more advantageous compared to thoracothomy (decrease of post surgery pains, decrease of recovery time and decrease of drugs consumption). Nevertheless, thoracoscopy needs specific materiels and nécessite un équipement spécifique and trained physicians. In France, only 1% of surgeries qu'en France, thoracoscopy represents less than 1% of lung cancer surgeries while it represents 30% of interventions in Japan.

Moreover, this technic needs that nodes was well localized. For this, radiologists use CT-guided hook wire localization of these lung nodes before surgery.

According to the litterature, this localization technic is efficient (Chen et al, 2011).

The hook wire laying is delicate. It can lead secondaries effects as pneumothorax, dislodgement of the hook wire before and after surgery. The success rate of hook wire fixation in lung near of the node is primary.

The main objective of our study is to assess the success rate localization of node in surgery piece, that is to verify if the hook wire have allowed to localize the lung node in surgery piece. This implies that:

* the hook wire was well CT-guided in the lung
* the hook wire did not present a dislodgment before or during surgery
* the hook wire is near of the node to be removed Among secondaries objectives, the investigators will assess the safety and possible complications which could occur. The investigators will also measure the distance between hook wire and center of the node

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patient with suspect lung node, needed surgery
* Signed consent

Exclusion Criteria:

* Too deep node
* Severe co-morbidities : respiratory insufficiency, cardiac insufficiency
* Major emphysema
* Patient with only one lung
* Pregnant women
* Breastfeeding women
* Patient with cognitive and psychiatric troubles

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Nodule detection in surgery piece (success rate) | At surgery

SECONDARY OUTCOMES:
Nodule detection under scanner | After patient inclusion, at scan realisation, before surgery. This detection will be realised up to 4 weeks after inclusion.
Adverse events assessment graded with NCI -CTCAE v4.0 | Before and after surgery, up to 4 weeks after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Jean Perrin, Clermont-Ferrand, France